CLINICAL TRIAL: NCT03229421
Title: Survey of Symptoms and Dermatologic Characterization Associated With Zika Virus
Brief Title: Dermatologic Manifestations of Zika Virus
Acronym: DMZV
Status: Withdrawn | Type: Observational
Why Stopped: Unable to enroll eligible participants
Sponsor: Northwestern University (Other)
Collaborators: Pontificia Universidad Catolica Madre y Maestra (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Principal Investigator, Northwestern University
Other Study IDs: STU00205325
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Zika Virus Symptoms and the Associated Exanthema
Keywords: Zika Virus
MeSH Terms: conditions — Zika Virus Infection | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — 18 question symptom assessment tool including non-identifying demographic information questions.

SUMMARY:
The purpose of this study is to determine whether any diagnostic patterns exist in the symptom presentation of Zika Virus.

DETAILED DESCRIPTION:
The study has both retrospective and prospective components. The retrospective review includes medical records with laboratory confirmed Zika Virus diagnosis and the prospective component will enroll adults presenting with febrile illness and rash and ask them to complete a survey about their symptoms. Diagnostic testing will be completed to confirm infection source.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older presenting with febrile illness and rash

Exclusion Criteria:

* Patients aged 17 years or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 y/o with confirmed zika virus diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of days with specific symptoms | 20 minutes
  Number of days reported experiencing specific symptoms due to Zika Virus infection and and associated characteristics such as location and intensity

SECONDARY OUTCOMES:
Frequency measures of initial clinical presentations | 20 minutes
  Frequency of reported symptoms at initial clinical presentation.

CONTACTS AND LOCATIONS:
Overall Officials: Roopal V. Kundu, MD, Principal Investigator — Northwestern University
Locations (1):
- Pontificia Universidad Catolica Madre y Maestra, Departamento de Medicina, Santo Domingo, Illinois, Dominican Republic

IPD SHARING:
Plan to Share IPD: No